CLINICAL TRIAL: NCT01387711
Title: A Phase I, Single-centre, Open Label, Within-subject Comparison Trial to Explore the Biological Effects of PEP005 (Ingenol Mebutate) Gel, 0.05%, Applied Once Daily for 2 Consecutive Days in Patients With Actinic Keratosis on the Upper Extremity
Brief Title: PEP005 Gel - Biological Effects in Actinic Keratosis Assessed by Histology
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LP0041-02
Record Dates: First submitted 2011-07-01; First posted 2011-07-04 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2016-12

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ingenol mebutate (Experimental): PEP gel 0.05% once daily exposure
  Interventions: Drug: PEP005 (Ingenol mebutat Gel, 0.05 %)

INTERVENTIONS:
Drug: PEP005 (Ingenol mebutat Gel, 0.05 %) — All eligible patients will receive PEP005 Gel, 0.05 %, on two consecutive days to both the AK Treatment Area and the Normal Skin Treatment Area

SUMMARY:
This trial will be conducted to explore the biological effects in the skin following treatment with PEP005 Gel, 0.05% administered for two consecutive days, assessed by histology.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients at least 18 years of age
2. Patients with AK lesions within a contiguous 25 cm2 area on the upper extremity
3. Patients with a 25 cm2 area of normal skin on the upper inner arm
4. Female subjects must be of either non-childbearing potential or childbearing potential, provided there is a confirmed negative urine pregnancy test prior to exposure, to rule out pregnancy
5. Female subjects of childbearing potential must be willing to consent to using high effective methods of contraception
6. Ability to follow study instructions and likely to complete all study requirements
7. Obtained written informed consent prior to any study-related procedures

Exclusion Criteria:

1. Location of the selected treatment areas within 5 cm of an incompletely healed wound within 10 cm of a suspected basal cell carcinoma (BCC) or squamous cell carcinoma (SCC)
2. History or evidence of skin conditions other than the study indication that would interfere with evaluation of the study medication
3. Clinical diagnosis/history or evidence of any medical condition that would expose a subject to an undue risk of a significant AE or interfere with assessments of safety, as determined by Investigator clinical judgment.
4. Anticipated need for in-patient hospitalisation or in-patient surgery during the study period.
5. Current participation in any other interventional clinical trial
6. Subjects who have received treatment with any non-marketed drug product within the last two months
7. Subject known or, in the opinion of the investigator, is unlikely to comply with the Clinical Study Protocol
8. Females who are pregnant, of child-bearing potential and wishing to become pregnant during the trial, or are breast feeding
9. Undergone cosmetic or therapeutic procedures within 2 cm of the selected treatment areas in the 2 weeks prior to the screening visit
10. Use of acid-containing therapeutic products within 2 cm of the selected treatment areas in the 2 weeks prior to the screening visit
11. Use of topical salves/topical steroids: within 2 cm of the selected treatment areas in the 2 weeks prior to the screening visit
12. Treatment with immunomodulators, cytotoxic drugs or interferon/interferon inducers, systemic medications that suppress the immune system or UVB in the last 4 weeks
13. Treatment with 5-FU, imiquimod, diclofenac, or photodynamic therapy: within 2 cm of the selected treatment areas within 8 weeks prior to any screening visit
14. Use of systemic retinoids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Leukocytes Infiltration and degree of necrosis of the AK lesion and skin | From baseline until day 3
  Degree of skin infiltration of leukocytes and necrosis of the epidermis and dermis in the AK biopsies from Day 1, Day 2, and Day 3

SECONDARY OUTCOMES:
Biological effects in the skin | from baseline till day day 3
  * Leukocytes Infiltration
  * Degree of skin infiltration of leukocytes
  * Necrosis
  * Haemorrhage
  * Immune cell activation
  * Apoptosis
  * Endothelium activation
  * RNA expression
  * Drug Transporter
  Number of participants with changes in normal skin and AK lesion biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Schön, MD, Principal Investigator — Universitätsmedizin Göttingen, Georg-August-Universität
Locations (1):
- Universitätsmedizin Göttingen, Georg-August-Universität, Göttingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Emmert S, Haenssle HA, Zibert JR, Schon M, Hald A, Hansen MH, Litman T, Schon MP. Tumor-Preferential Induction of Immune Responses and Epidermal Cell Death in Actinic Keratoses by Ingenol Mebutate. PLoS One. 2016 Sep 9;11(9):e0160096. doi: 10.1371/journal.pone.0160096. eCollection 2016. PMID 27612149
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en